CLINICAL TRIAL: NCT01720225
Title: Phase II Randomized Study of Lower Doses of Decitabine (DAC; 20 mg/m2 IV Daily for 3 Days Every Month) Versus Azacitidine (AZA; 75 mg/m2 SC/IV Daily for 3 Days Every Month) in Myelodysplastic Syndrome (MDS) Patients With Low and Intermediate-1 Risk Disease
Brief Title: Decitabine Versus Azacitidine in Myelodysplastic Syndrome Patients With Low and Intermediate-1 Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0507; NCI-2012-02215 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndromes; MDS; Low and Intermediate-1 Risk Disease; Decitabine; DAC; Dacogen; Azacitidine; AZA; 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Decitabine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decitabine (Experimental): Patients randomized to receive Decitabine 20 mg/m2 by vein daily for 3 days (days 1-3) every 28 days.
  Interventions: Drug: Decitabine
- Azacitidine (Experimental): Patients randomized to receive Azacitidine 75 mg/m2 subcutaneously or by vein daily for 3 days (days 1-3) every 28 days.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Decitabine — 20 mg/m2 by vein daily for 3 days (days 1-3) every 28 days.
  Other Names: DAC; Dacogen
  Arms: Decitabine
Drug: Azacitidine — 75 mg/m2 subcutaneously or by vein daily for 3 days (days 1-3) every 28 days.
  Other Names: AZA; 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Azacitidine

SUMMARY:
The goal of this clinical research study is to compare how two different drugs, decitabine and azacitidine, when given on a shorter than standard dosing schedule can help to control MDS. The safety of the drugs will also be studied.

Decitabine is designed to damage the DNA (the genetic material) of cells, which may cause cancer cells to die.

Azacitidine is designed to block certain proteins in cancer cells whose job is to stop the function of the tumor-fighting proteins. By blocking the "bad" proteins, the tumor-fighting genes may be able to work better. This could cause the cancer cells to die.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups:

* If you are in Group 1, you will receive decitabine by vein over about 1 hour.
* If you are in Group 2, you will receive azacitidine either as an injection under your skin or through a vein. If by vein, the infusion will take about an hour.

At first, there will be an equal chance of being assigned to either group. However, as the study goes on and more information becomes available, the chance of being assigned to the group that has shown the most effectiveness will increase. However, once you are already enrolled and assigned to a group, you will not be eligible to change groups.

Study Drug Administration:

Each cycle is 28 days.

You will receive the study drug on Days 1-3 of every cycle and you will receive at least 2 cycles of study drug.

Study Visits:

Every 7-14 days, blood (about 2 tablespoons) will be drawn for routine tests.

At the end of Cycle 2, you will have a bone marrow biopsy and/or aspirate to check the status of the disease. This will then be repeated every 2-4 cycles until any point that the disease appears to have responded to the study drug, then as often as the study doctor thinks is necessary. To collect a bone marrow biopsy/aspirate, an area of the hip bone is numbed with anesthetic, and a small amount of bone and/or bone marrow is withdrawn through a large needle.

After Cycle 3:

If the study doctor decides it is acceptable, you may be allowed to receive treatment from your local cancer doctor. However, you have to return to Houston at least every 3 months for your study visits.

The frequency of the visits will depend on what the doctor thinks is in your best interest.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Follow-Up Visits:

One (1) time every 3 months after your last dose of study drug, you will return to the clinic for a bone marrow aspiration to check the status of the disease.

Other Information:

You may be given other drugs to help prevent side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

This is an investigational study. Decitabine and Azacitidine are both FDA approved and commercially available for use in patients with MDS.

Up to 120 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an Institutional Review Board (IRB)-approved informed consent document.
2. Age >/= than18 years
3. de novo or secondary International Prostate Symptom Score (IPSS) low- or intermediate-1 - risk MDS, including CMML
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 3 at study entry.
5. Organ function as defined: Serum creatinine </= 3 x Upper Limit of Normal (ULN), Total bilirubin </= 2 x ULN, Alanine transaminase (ALT) (SGPT) </= 2 x ULN
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days and will also need to use contraceptives. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.

Exclusion Criteria:

1. Breast feeding females
2. Prior therapy with decitabine or azacitidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sasaki K, Jabbour E, Montalban-Bravo G, Darbaniyan F, Do KA, Class C, Short NJ, Kanagal-Shamana R, Kadia T, Borthakur G, Pemmaraju N, Cortes J, Ravandi F, Alvarado Y, Chien K, Komrokji R, Sekeres MA, Steensma DP, DeZern A, Roboz G, Soltysiak K, Yang H, Kantarjian HM, Garcia-Manero G. Low-Dose Decitabine versus Low-Dose Azacitidine in Lower-Risk MDS. NEJM Evid. 2022 Oct;1(10):EVIDoa2200034. doi: 10.1056/EVIDoa2200034. Epub 2022 Aug 9. PMID 38319837
- [Derived] Jabbour E, Short NJ, Montalban-Bravo G, Huang X, Bueso-Ramos C, Qiao W, Yang H, Zhao C, Kadia T, Borthakur G, Pemmaraju N, Sasaki K, Estrov Z, Cortes J, Ravandi F, Alvarado Y, Komrokji R, Sekeres MA, Steensma DP, DeZern A, Roboz G, Kantarjian H, Garcia-Manero G. Randomized phase 2 study of low-dose decitabine vs low-dose azacitidine in lower-risk MDS and MDS/MPN. Blood. 2017 Sep 28;130(13):1514-1522. doi: 10.1182/blood-2017-06-788497. Epub 2017 Aug 3. PMID 28774880
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2012 to February 2016
Period: Overall Study
Arm/Group | Decitabine | Azacitidine
Started | 73 | 40
Completed | 70 | 39
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Did not complete 2 cycles of therapy | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine | Azacitidine | Total
Number analyzed (Participants) | 73 | 40 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 12 | 38
  >=65 years | 47 | 28 | 75
Age, Continuous [Median (Full Range); unit: years] | 70 [44 to 88] | 70 [53 to 84] | 70 [44 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 49 | 24 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 71 | 39 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 40 | 113

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Overall Response = complete remission (CR) + partial remission (PR) + marrow CR (mCR) + hematologic improvement (HI). CR is normalization of peripheral blood and bone marrow with <5% bone marrow blasts, a peripheral blood granulocyte count > (1.0 x 10^9/L, and platelet count > 100 x 10^9/L). PR is same as CR except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment. Marrow CR is blasts </= 5% and decreased by >/=50% from baseline. HI is platelets increase by 50% and to above 30 x 10^9/L untransfused (if lower than that pre-therapy; or hemoglobin increase by 2 g/dl; or transfusion independent; or splenomegaly reduction by > 50%; or monocytosis reduction by > 50% if pretreatment > 5 X1 0^9/L.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine | Azacitidine
Number analyzed (Participants) | 70 | 39
Participants | 49 | 19

2. Secondary Outcome: Number of Participants Who Became Transfusion Independent
Description: Participants who were transfusion dependent at baseline prior to starting therapy on the Decitabine or Azacitidine arm will be analyzed for transfusion independence. Transfusion independence defined as being transfusion-free for ≥8 consecutive weeks between the first dose and study treatment discontinuation.
Time Frame: 8 weeks
Population: Participants analyzed for Transfusion Independence must have been transfusion dependent at baseline. Thirty-seven participants in the Decitabine arm and nineteen participants in the Azacitidine arm where transfusion dependent prior to treatment on this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine | Azacitidine
Number analyzed (Participants) | 37 | 19
Participants | 12 | 3

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Arm/Group | Decitabine | Azacitidine
All-Cause Mortality (participants affected / at risk) | 7/73 | 2/40
Serious Adverse Events (participants affected / at risk) | 32/73 | 14/40
Other Adverse Events (participants affected / at risk) | 20/73 | 16/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=73) | Azacitidine (N=40)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Altered Mental Status (Nervous system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 1 (1) | 0 (0)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (3) | 0 (0)
Food Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Groin Abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 2 (3) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Joint Infection (Infections and infestations) | 1 (1) | 0 (0)
Left plerual effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leg Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 3 (3) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 9 (17) | 2 (2)
Otitis Externa (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pain Abdominal Abcess (General disorders) | 1 (1) | 0 (0)
Pain Right Extremity (General disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 1 (4)
Right atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal Hermorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Right Hip Pain (General disorders) | 0 (0) | 1 (1)
Salmonella Bactremia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sialadenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small Intestine Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Submandibular Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Syncopal episode (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Vaginal Fistual (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=73) | Azacitidine (N=40)
Nausea (Gastrointestinal disorders) | 11 (11) | 6 (6)
Fatigue (General disorders) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT01720225/Prot_SAP_000.pdf